CLINICAL TRIAL: NCT04408352
Title: Selective Bladder Denervation Using RF Energy for the Treatment of UUI
Brief Title: RF Ablation of the Trigone for the Treatment of UUI
Acronym: TRANSFORM
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: for business planning purposes only, and is not related to any safety or performance issues identified during the study
Sponsor: Hologic, Inc. (Industry)
Collaborators: NAMSA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1360-001
Record Dates: First submitted 2020-05-26; First posted 2020-05-29 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Urgent Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to either the treatment with the Hologic trigone RF ablation device or a sham procedure. Randomization will occur in a 2:1 fashion (treatment: sham) meaning approximately 150 subjects will be treated with the Hologic trigone RF ablation device and 75 control subjects treated with the sham procedure. Randomization will be stratified by site.
Who Masked: Participant, Outcomes Assessor
Masking Description: The device shall be assembled and maintained in a sterile environment outside the view of the subject during procedure preparation and treatment. The treating investigator, applicable nursing and site staff, and any representatives supporting the procedure should refrain from discussing the device or treatment assignment during the procedure and applicable follow-up visits. The sham procedure will mimic the Hologic trigone RF ablation device procedure to maintain subject blinding and provide the most accurate assessment of control data while minimizing risk to the subject. Energy will not be delivered to the tissue when each sham "ablation" is started.To be comparable to the Hologic trigone RF ablation device procedure, the simulated ablation procedure will need to be repeated as many times as necessary to cover the area of the trigone as is done in the treatment arm.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- RF Trigone Ablation Treatment Arm (Active Comparator): A compatible standard cystoscopy lens (30°) will be inserted into the Hologic trigone RF Device. The bladder will be emptied of urine and saline infused into the bladder to allow adequate visualization and working space. Ablations at the trigone will be created using the Hologic trigone RF ablation device together with the compatible standard commercially available RF cannula and generator. It is expected that a subject would receive between 4-6 ablations to completely treat the appropriate area of the trigone. At the completion of the procedure, 200 ml of saline is instilled into the bladder to allow for assessment of voiding function prior to discharge.
  Interventions: Device: selective bladder denervation using RF energy
- RF Trigone Ablation Sham Arm (Sham Comparator): The sham procedure will mimic the Hologic trigone RF ablation device procedure to maintain subject blinding and provide the most accurate assessment of control data while minimizing risk to the subject.
  The bladder will be emptied of urine and saline infused into the bladder to allow adequate visualization and working space. Suction will be applied to the bladder wall and the cannulas (needles) will be introduced into the bladder wall. Energy will not be delivered to the tissue when each sham "ablation" is started. In order to maintain blinding of the subject, the typical sounds that Hologic trigone RF ablation device makes during actual ablation/fulguration will be replicated. The simulated ablation procedure will be repeated as many times as necessary to cover the area of the trigone. 4 to 6 sham "ablations" would be required. At the completion of the procedure, 200ml of saline is instilled into the bladder to allow for assessment of voiding function prior to discharge.
  Interventions: Device: selective bladder denervation using RF energy

INTERVENTIONS:
Device: selective bladder denervation using RF energy — RF ablation of the trigone for the treatment of UUI

SUMMARY:
The primary objective of this pivotal study is to collect data on the safety and effectiveness of the Hologic trigone RF ablation device to reduce urgency urinary incontinence. Up to 325 subjects will be enrolled with 225 randomized (2:1) and treated at up to 35 sites in the U.S. Additional sites in Canada, Australia, Europe, and other countries may also be considered. Sites outside of the U.S. cannot randomize more than 25% of subjects.

DETAILED DESCRIPTION:
Up to 325 subjects who meet all inclusion and none of the exclusion criteria will be enrolled and up to 225 subjects will be randomized. Subjects will be randomized to either an active arm that includes treatment with the Hologic trigone RF ablation device, or a control arm who receive a sham procedure. With a 2:1 randomization, approximately 150 subjects will be treated with the Hologic trigone RF ablation device (treatment group) and 75 sham subjects treated with the sham procedure.

Subjects will be blinded to their randomized treatment; however, due to the nature of the procedure, the treating investigator cannot be blinded to individual randomization assignments.

Subjects who are randomized to the treatment arm will be followed at 2 weeks, 1 month, 3, 6, and 12 months and every 6 months thereafter. Subjects randomized to the sham arm will be followed through the 6-month visit. Follow up of all other subjects (cross-over and treatment arm) will conclude when the last subject in randomized treatment arm reaches their 12-month visit, is withdrawn, or is determined lost to follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Non-pregnant, non-lactating female NOTE: Females who are of childbearing potential must have had a negative pregnancy test <7 days prior to procedure and must be using medically accepted contraception or have a monogamous relationship with a partner who has undergone sterilization.
2. Subject is ≥18 years of age
3. Subject has a history of idiopathic UUI for ≥ 6 months
4. Subject is willing to provide Informed Consent, is geographically stable, has the cognitive ability to complete the 3-day bladder diary and comply with the required diary, follow up visits and testing schedule requirements
5. Ambulatory and able to use toilet without assistance
6. Post-void residual (PVR) ≤ 150 ml
7. Intolerant of, contraindicated for, or have failed drug therapy AND should not be on medications for their condition for at least 2 weeks prior
8. Predominance of urgency urinary incontinence in subjects with mixed incontinence (mix of both stress and urgency incontinence) NOTE: Predominance is defined as having at least 2/3rds or 67% of reported incontinence as urgency urinary incontinence on the 3-day bladder diary, and a higher percentage urgency urinary incontinence score as compared to the SUI score on the MESA-UIQ
9. Subject has not previously received, or did receive ≤ 100 units/intravesical treatment of Onabotulinum Toxin A (Botox®) for OAB and self-reports receiving benefit from Botox of normal durability (3-6 months), but discontinued or wishes to discontinue due to side effects, financial constraints, or required treatment regimen (e.g., treatment every 6 months)
10. ≥ 4 episodes of urgency urinary incontinence (UUI) over 3-day Bladder Diary (an average of 1.33 UUI episodes/day)

Exclusion Criteria:

1. Planning on becoming pregnant during the 36-month study period
2. Serum creatinine or BUN > twice the upper limit of normal within the last sixty days; Impaired renal function as measured by glomerular filtration rate (GFR) ≤ 65
3. Current bleeding disorder or coagulopathies
4. Neurological disease affecting bladder function such as multiple sclerosis, spinal cord injuries, myasthenia gravis, Charcot-Marie-Tooth disease
5. Subject has uncontrolled diabetes (HbA1C >8.5) documented in the last three months
6. Subject is a chronic corticosteroid user defined as daily continuous use within the last 30 days
7. Subject is critically ill or has a life expectancy <3 years
8. Investigator determines that subject is not a suitable candidate for participation in an investigational clinical research study
9. Post-surgical onset of de novo OAB
10. Current hydronephrosis or hydroureter
11. Patients with uninvestigated microhematuria
12. Impaired voiding dysfunction due to underactive bladder or bladder outflow obstruction
13. Current participation in any other interventional study. Participation in observational studies is permitted
14. Prior or current diagnosis of polyuria or has a screening 3-day bladder diary with 24-hour total volume of > 3000 ml
15. Urinary tract infection (UTI) that is not resolved or has not been treated with antibiotics for a minimum of 3 days at the time of procedure and has not been verified by a negative urinalysis
16. Subject reports having, or has a documented history of ≥ 2 urinary tract infections (UTIs) in the last 6 months, or ≥3 UTIs in the last 12 months prior to enrollment
17. Documented, spontaneous, unprovoked urinary retention requiring any type of catheterization within the last 6 months or retention in the past for which there was no diagnosis or definitive treatment
18. Anatomical conditions that, in the opinion of the investigator, would preclude the introduction and/or use of the device
19. Any prolapse at or beyond the hymen
20. Subject has been diagnosed (at any time) with bladder cancer, interstitial cystitis or chronic pelvic pain syndrome
21. Ureteral dysfunction, stricture or reflux including vesicoureteral reflux or a history of surgical treatment for vesicoureteral reflux
22. Any abnormality of the urinary tract including the bladder, ureters or kidneys such as but not limited to: hydroureter, hydronephrosis, ureteric reflux, Hutch diverticulum, ureterocele, duplex system, ectopic ureter, unilateral renal agenesis, ectopic kidney, cross fused ectopia, or megaureter
23. Any invasive or surgical intervention involving the kidneys, bladder, urethra, rectum or vaginal wall within the last 6 months (e.g., radiofrequency, implant, mid-urethral sling)
24. Prior history of surgical mesh in the anterior vaginal compartment to treat pelvic organ prolapse
25. History of complications with any transvaginal or mid-urethral implanted mesh
26. Prior abdominal, pelvic or vaginal surgery that may have modified the structure or location of the bladder, ureters or urinary vasculature such as bladder reconstruction, retroperitoneal dissection or cross-trigonal ureteral implantation, urinary tract fistula repair
27. Current use of OAB medications within the last 2 weeks
28. OAB symptoms previously treated with a single injection of >100 units of Onabotulinum Toxin A (Botox®)
29. OAB symptoms previously treated with Sacral Neuromodulation (SNM) and/or PTNS
30. Previous pelvic irradiation
31. Complete or total incontinence (i.e. the continuous or total loss of urinary control)
32. Any functional incontinence (incontinence caused by a physical or mental impairment that keeps a subject from reaching the bathroom in time to urinate)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study will enroll adult (≥18 years of age), female subjects with urgency urinary incontinence (UUI) who are found to be intolerant of, contraindicated for, or have failed drug therapy and are not on medications for their condition.
Enrollment: 225 (Estimated)
Dates: Start 2020-04-27 (Actual); Primary Completion 2030-02 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint | 6 months
  The proportion of UUI responders having a > 50% decrease in UUI episodes from baseline to 6-month follow-up as documented on the 3-day bladder diary.
Primary Safety Endpoint | 12 months
  All adverse events from randomized treatment through the close of the 12-month follow-up visit for subjects treated with the Hologic trigone RF ablation device.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Cypress Medical Research Center, LLC, Wichita, Kansas
  - Regional Urology, LLC, Shreveport, Louisiana
  - UPMC Magee Womens Hospital, Pittsburgh, Pennsylvania
  - Alleghany Health Network, Pittsburgh, Pennsylvania
  - Center for Pelvic Health, Franklin, Tennessee
  - Virginia Urology, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No